CLINICAL TRIAL: NCT06774274
Title: Analgesic Efficacy of Intravenous Ketamine as a Continuous Infusion vs PCA in the Management of Acute Postoperative Pain in Major Orthopedic Surgery: A Randomized Clinical Trial
Brief Title: Analgesic Efficacy of Intravenous Ketamine as a Continuous Infusion vs PCA in the Management of Acute Postoperative Pain in Major Orthopedic Surgery.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Hospital San Vicente Fundación (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36-2024
Record Dates: First submitted 2025-01-07; First posted 2025-01-14 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Opioid Use; Major Surgery
Keywords: postoperative pain; ketamine; patient controlled analgesia; continuous infusion; major surgery; pain; abdominal surgery; thoracic surgery; spine surgery; opioid; major orthopedic surgery
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: This trial will be a triple-blind, parallel-group, pragmatic, non-inferiority controlled clinical trial focused on pain management and superiority regarding opioid use, along with other secondary outcomes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treating Anesthesiologist: The anesthesiologist responsible for the case and intraoperative management will be blinded to the assigned intervention. The assignment will be carried out by another anesthesiologist who is not involved in the case. This external anesthesiologist will be present in the operating room, and after opening the envelope, will inform the nursing staff regarding which drug mixtures to prepare.
  Data Collection and Analysis Staff: Data will be collected during the hospital stay, up to three days, by two researchers. The researchers will be blinded to the assignment and will not have access to information about the prepared drug mixtures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine infusion (Active Comparator): Intravenous ketamine administered as a continuous infusion.
  Interventions: Drug: Ketamine infusion
- PCA Ketamine (Active Comparator): Intravenous ketamine administered along with opioid in a single saline bag using a Patient Controlled Analgesia pump
  Interventions: Drug: PCA Ketamine

INTERVENTIONS:
Drug: Ketamine infusion — A 10% ketamine solution will be prepared in a 250 cc bag of 0.9% saline (1 mg/cc) using 5 cc from a vial of ketamine that has a concentration of 50 mg/cc. The infusion will be initiated at the time of surgical site closure and will proceed as follows: a bolus of 0.35 cc/kg (equivalent to 0.35 mg/kg) will be administered, followed by a continuous infusion of 0.1 cc/kg/h (equivalent to 0.1 mg/kg/h) for up to 48 hours postoperatively.
  Patients in this group will have access to a PCA pump with morphine for analgesic rescue and to monitor daily opioid consumption.
  Arms: Ketamine infusion
Drug: PCA Ketamine — A mixture of 5% ketamine and 5% morphine will be prepared in a 100 cc bag of 0.9% saline. This will be achieved by using 1 cc of a ketamine vial (50 mg/cc) and 5 cc of a morphine ampule (10 mg/cc). This results in a final concentration of 0.5 mg of ketamine and 0.5 mg of morphine per cc in the 100 cc saline bag.
  The pump settings will be configured as follows:
  * PCA (Patient-Controlled Analgesia) dose: 2 cc (which delivers 1 mg of ketamine and 1 mg of morphine)
  * Lockout interval: 6 minutes
  * Maximum dose limit: 15 doses over a 4-hour period
  The pump will be available for patient use for up to 48 hours postoperatively.
  Other Names: Ketamine PCA
  Arms: PCA Ketamine

SUMMARY:
The goal of this clinical trial is to determine whether treating pain after surgery with ketamine is more effective when administered intravenously as a continuous infusion or through a patient-controlled analgesia (PCA) pump. This study focuses on adult volunteers following major orthopedic surgery. We have two main questions to address:

* Is a continuous intravenous infusion of ketamine as effective as ketamine administered through a PCA pump for managing pain after major orthopedic surgery.
* Does a continuous intravenous infusion of ketamine result in lower opioid requirements compared to ketamine delivered through a PCA pump for pain management after major orthopedic surgery?

Participants will be divided into two groups. One group will receive ketamine via continuous infusion, while the other will receive it through a PCA pump. Both groups will also receive a placebo (a substance that looks like the drug but contains no active ingredients), ensuring that neither group knows whether they are receiving ketamine through the PCA pump (which always contains a painkiller) or as a continuous infusion.

Participants will be assigned to one of the two groups and will receive their assigned treatment for 48 hours while hospitalized. Researchers will visit participants during their first three days in the hospital to assess their pain levels and monitor for any side effects.

DETAILED DESCRIPTION:
Managing postoperative pain is a primary concern for patients undergoing major surgery, especially in major orthopedic surgery. Effective pain management is crucial, as uncontrolled postoperative pain can lead to prolonged hospital stays, decreased patient satisfaction, and various complications, including pulmonary and gastrointestinal issues.

Current pain management strategies emphasize multimodal analgesia, which involves using multiple medications with different mechanisms of action to minimize side effects. Ketamine has been investigated in this context and has been found effective for treating postoperative pain following major surgeries while reducing the need for opioids. However, there is still some uncertainty regarding the optimal method for administering ketamine after surgery. The aim of this trial is to compare the effectiveness of intravenous ketamine in terms of pain control, measured by numerical pain scores, and opioid consumption within the first 24 hours postoperatively using two different strategies: continuous infusion versus patient-controlled analgesia (PCA) in adults undergoing non-cardiac surgery.

For this research, two hypotheses are proposed, as the objective involves two types of outcomes related to the analgesic effectiveness of intravenous ketamine: pain measured by a numerical pain scale and opioid consumption equivalent to oral morphine.

Based on data from previous studies, it is highly likely that continuous ketamine infusion will provide similar pain control efficacy at 24 hours compared to PCA ketamine. However, the data suggests that continuous infusion may result in lower opioid consumption than PCA. Therefore, the hypotheses are as follows:

**First Hypothesis** Continuous ketamine infusion is not inferior to PCA ketamine for pain control, as measured by a numerical pain scale at 24 hours postoperatively in patients undergoing major orthopedic surgery with a high risk of severe acute pain.

**Second Hypothesis** Continuous ketamine infusion is superior to PCA ketamine in reducing opioid consumption at 24 hours postoperatively in patients undergoing major orthopedic surgery at high risk of severe acute pain.

This trial will be a triple-blind, parallel-group, pragmatic, non-inferiority controlled clinical trial focused on pain management and superiority regarding opioid use, along with other secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Elective major orthopedic surgery.
* ASA (American Association of Anesthesiology) classification 1, 2 or 3.

Exclusion Criteria:

* Patients with a diagnosis of perioperative kidney injury or hepatic failure
* Patients with active cardiac conditions
* Patients with any cognitive impairment that disables the patient from operating the PCA pump or impedes the postoperative interview
* Patients with scheduled ICU admission with invasive ventilatory support
* Patients with known hypersensitivity to opioid medications
* Patients with past medical history of severe adverse reactions to opioids or ketamine.
* Pregnant patients
* Patients undergoing continuous regional anesthetic techniques including peripheral nerve catheters or continuous epidural catheters
* Patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours after surgery
  Visual Analog Scale (VAS) for dynamic (during movement) pain. The VAS for pain is a unidimensional measure of pain intensity in adults.The pain VAS is a continuous visual scale from 0 to 100 mm, with 0 mm representing "no pain" and 100 mm representing maximum pain (e.g. "worst pain imaginable").
Postoperative opioid use | 24 hours after surgery
  Daily opioid use expressed in morphine equivalents (morphine equivalent daily dose MEDD)

SECONDARY OUTCOMES:
Dynamic and rest postoperative pain | 12, 24, 48, and 72 hours after surgery
  Visual Analog Scale (VAS) for dynamic and rest postoperative pain . The VAS for pain is a unidimensional measure of pain intensity in adults.The pain VAS is a continuous visual scale from 0 to 100 mm, with 0 mm representing "no pain" and 100 mm representing maximum pain (e.g. "worst pain imaginable")
Postoperative opioid use | 48 and 72 hours after surgery
  Daily opioid use expressed in morphine equivalents (morphine equivalent daily dose MEDD)
Time to ambulation | 72 hours after surgery
  Time measured in days for the patient to begin ambulation after surgery.
Hospital stay | From date of randomization until the date day of discharge or date of death from any cause, whichever came first, assessed up to 36 months
  Days of hospital stay
Postoperative nausea and vomiting | 24 hours after surgery
  Proportion of patients with at least one episode of nausea or vomiting after surgery
Respiratory depression | 72 hours after surgery
  Proportion of patients with any episode of respiratory rate <8 breaths per minute accompanied by supplemental oxygen requirement higher than a simple nasal cannula; or the requirement of facial mask ventilation or tracheal intubation; or requirement of naloxone reversal
Oversedation | 2, 12, 24, 48, and 72 hours after surgery
  Proportion of patients with any episode of sedation measured as a level 4 or higher using Ramsay's sedation scale
Psychomimetic symptoms | 72 hours after surgery
  Proportion of patients with at least one of the following symptoms:
  * Hallucinations: Defined as any tactile, visual, auditory, or sensory experience in the absence of an appropriate stimulus, referred by the patient as real
  * Nightmares: Defined as any vivid dream with a negative or dysphoric emotional content
Delirium | 72 hours after surgery
  Proportion of patients diagnosed with delirium using the Confusion Assessment Method scale
Hemodynamic measurements - Arterial pressure | 2, 12, 24, 48, and 72 hours after surgery
  Systolic, diastolic, and mean arterial pressure in mmHg.
Hemodynamic measurements - Heart rate | 2, 12, 24, 48, and 72 hours after surgery
  Heart rate in beats per minute.
Urinary retention | 72 hours after surgery
  Proportion of patients with any event of impossibility for spontaneous micturition reported by the patient requiring physical measures or urinary catheter insertion for resolution
Pruritus | 72 hours after surgery
  Proportion of patients reporting any episode of itching in any body region
Time to first bowel movement | 72 hours after surgery
  Measured in time to initiation of the first passing of stool or flatus

CONTACTS AND LOCATIONS:
Overall Officials: Fabian D Casas, Professor, Study Chair — Universidad de Antioquia
Locations (1):
- St. Vincent's Foundation University Hospital, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No
It was not approved by our Institutional Research Board.

REFERENCES:
- [Background] Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE, Dixon-Woods M, McCulloch P, Wyatt JC, Chan AW, Michie S. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. BMJ. 2014 Mar 7;348:g1687. doi: 10.1136/bmj.g1687. PMID 24609605
- [Background] Jouguelet-Lacoste J, La Colla L, Schilling D, Chelly JE. The use of intravenous infusion or single dose of low-dose ketamine for postoperative analgesia: a review of the current literature. Pain Med. 2015 Feb;16(2):383-403. doi: 10.1111/pme.12619. Epub 2014 Dec 19. PMID 25530168
- [Background] Laskowski K, Stirling A, McKay WP, Lim HJ. A systematic review of intravenous ketamine for postoperative analgesia. Can J Anaesth. 2011 Oct;58(10):911-23. doi: 10.1007/s12630-011-9560-0. Epub 2011 Jul 20. PMID 21773855
- [Background] Waelkens P, Alsabbagh E, Sauter A, Joshi GP, Beloeil H; PROSPECT Working group * * of the European Society of Regional Anaesthesia and Pain therapy (ESRA). Pain management after complex spine surgery: A systematic review and procedure-specific postoperative pain management recommendations. Eur J Anaesthesiol. 2021 Sep 1;38(9):985-994. doi: 10.1097/EJA.0000000000001448. PMID 34397527
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Vadeghani AT, Grant M, Forget P. Perioperative pain management interventions in opioid user patients: an overview of reviews. BMC Anesthesiol. 2024 Sep 5;24(1):310. doi: 10.1186/s12871-024-02703-6. PMID 39237892
- [Background] Meyer-Friessem CH, Lipke E, Weibel S, Kranke P, Reichl S, Pogatzki-Zahn EM, Zahn PK, Schnabel A. Perioperative ketamine for postoperative pain management in patients with preoperative opioid intake: A systematic review and meta-analysis. J Clin Anesth. 2022 Jun;78:110652. doi: 10.1016/j.jclinane.2022.110652. Epub 2022 Jan 19. PMID 35065394
- [Background] Xu L, Xu S, Zhang Y, Huang Y. Effects of anesthetic adjunctive agents on postoperative cognitive dysfunction in elderly patients undergoing noncardiac surgery: A Bayesian network meta-analysis. Brain Behav. 2023 Aug;13(8):e3149. doi: 10.1002/brb3.3149. Epub 2023 Jul 11. PMID 37431799
- [Background] Sun W, Zhou Y, Wang J, Fu Y, Fan J, Cui Y, Wu Y, Wang L, Yu Y, Han R. Effects of Ketamine on Chronic Postsurgical Pain in Patients Undergoing Surgery: A Systematic Review and Meta-analysis. Pain Physician. 2023 May;26(3):E111-E122. PMID 37192226
- [Background] Aguirre-Cadavid LF, Ramírez-Luján CD, Casas-Arroyave FD, Calle-Cadavid E, Camelo-Rincón JE, Cadavid-Puentes AM. Psychomimetic Effects of Low-Dose Ketamine Infusions in Postoperative Pain: A Cohort Study.
- [Background] Cadavid AM, Casas FD, Camelo JE, Tovar A, Ramirez CD, Calle E, Visbal K. Effect of Analgesic Low-Dose Ketamine Infusions on the Cardiovascular Response: A Retrospective Analysis. Pain Physician. 2023 Sep;26(5):495-502. PMID 37774188
- [Background] Cadavid-Puentes AM, Camelo Rincón JE, Casas Arroyave FD, Chávez Lasso EF, Leyton Ortega M, Tovar Gutiérrez A. Hemodynamic response to sub-anesthetic doses of ketamine for postoperative pain: systematic review. Colomb J Anesthesiol. Available since february 12, 2024 52(2).
- [Background] Zhou JY, Hamilton P, Macres S, Pena M, Tang S. Update on Ketamine. Adv Anesth. 2020 Dec;38:97-113. doi: 10.1016/j.aan.2020.07.005. Epub 2020 Sep 14. No abstract available. PMID 34106842
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Hannon CP, Fillingham YA, Gililland JM, Sporer SM, Casambre FD, Verity TJ, Woznica A, Nelson N, Hamilton WG, Della Valle CJ. A Systematic Review of the Efficacy and Safety of Ketamine in Total Joint Arthroplasty. J Arthroplasty. 2023 Apr;38(4):763-768.e2. doi: 10.1016/j.arth.2022.10.037. Epub 2022 Oct 31. PMID 36328104
- [Background] Zhou L, Yang H, Hai Y, Cheng Y. Perioperative Low-Dose Ketamine for Postoperative Pain Management in Spine Surgery: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Pain Res Manag. 2022 Mar 31;2022:1507097. doi: 10.1155/2022/1507097. eCollection 2022. PMID 35401887
- [Background] Pendi A, Field R, Farhan SD, Eichler M, Bederman SS. Perioperative Ketamine for Analgesia in Spine Surgery: A Meta-analysis of Randomized Controlled Trials. Spine (Phila Pa 1976). 2018 Mar 1;43(5):E299-E307. doi: 10.1097/BRS.0000000000002318. PMID 28700455
- [Background] Terracina S, Robba C, Prete A, Sergi PG, Bilotta F. Prevention and Treatment of Postoperative Pain after Lumbar Spine Procedures: A Systematic Review. Pain Pract. 2018 Sep;18(7):925-945. doi: 10.1111/papr.12684. Epub 2018 Mar 25. PMID 29393998
- [Background] Zhaksylyk A, Abdildin YG, Sultangazin S, Zhumakanova A, Viderman D. The impact of ketamine on pain-related outcomes after thoracotomy: a systematic review with meta-analysis of randomized controlled trials. Front Med (Lausanne). 2024 Jun 11;11:1394219. doi: 10.3389/fmed.2024.1394219. eCollection 2024. PMID 38919936
- [Background] Akram U, Nadeem ZA, Ashfaq H, Fatima E, Ashraf H, Raza MA, Ahmed S, Nadeem A, Rehman S, Ahmad MH. Intraoperative ketamine and pain after video-assisted thoracoscopic surgery (VATS): A systematic review and meta-analysis. Anaesth Crit Care Pain Med. 2024 Dec;43(6):101444. doi: 10.1016/j.accpm.2024.101444. Epub 2024 Oct 16. PMID 39419346
- [Background] Brinck EC, Tiippana E, Heesen M, Bell RF, Straube S, Moore RA, Kontinen V. Perioperative intravenous ketamine for acute postoperative pain in adults. Cochrane Database Syst Rev. 2018 Dec 20;12(12):CD012033. doi: 10.1002/14651858.CD012033.pub4. PMID 30570761
- [Background] Garcia-Henares JF, Moral-Munoz JA, Salazar A, Del Pozo E. Effects of Ketamine on Postoperative Pain After Remifentanil-Based Anesthesia for Major and Minor Surgery in Adults: A Systematic Review and Meta-Analysis. Front Pharmacol. 2018 Aug 17;9:921. doi: 10.3389/fphar.2018.00921. eCollection 2018. PMID 30174603
- [Background] Wang L, Johnston B, Kaushal A, Cheng D, Zhu F, Martin J. Ketamine added to morphine or hydromorphone patient-controlled analgesia for acute postoperative pain in adults: a systematic review and meta-analysis of randomized trials. Can J Anaesth. 2016 Mar;63(3):311-25. doi: 10.1007/s12630-015-0551-4. Epub 2015 Dec 10. PMID 26659198
- [Background] Assouline B, Tramer MR, Kreienbuhl L, Elia N. Benefit and harm of adding ketamine to an opioid in a patient-controlled analgesia device for the control of postoperative pain: systematic review and meta-analyses of randomized controlled trials with trial sequential analyses. Pain. 2016 Dec;157(12):2854-2864. doi: 10.1097/j.pain.0000000000000705. PMID 27780181
- [Background] Levy N, Quinlan J, El-Boghdadly K, Fawcett WJ, Agarwal V, Bastable RB, Cox FJ, de Boer HD, Dowdy SC, Hattingh K, Knaggs RD, Mariano ER, Pelosi P, Scott MJ, Lobo DN, Macintyre PE. An international multidisciplinary consensus statement on the prevention of opioid-related harm in adult surgical patients. Anaesthesia. 2021 Apr;76(4):520-536. doi: 10.1111/anae.15262. Epub 2020 Oct 7. PMID 33027841
- [Background] McNicol ED, Ferguson MC, Hudcova J. Patient controlled opioid analgesia versus non-patient controlled opioid analgesia for postoperative pain. Cochrane Database Syst Rev. 2015 Jun 2;2015(6):CD003348. doi: 10.1002/14651858.CD003348.pub3. PMID 26035341
- [Background] Nardi-Hiebl S, Eberhart LHJ, Gehling M, Koch T, Schlesinger T, Kranke P. Quo Vadis PCA? A Review on Current Concepts, Economic Considerations, Patient-Related Aspects, and Future Development with respect to Patient-Controlled Analgesia. Anesthesiol Res Pract. 2020 Feb 13;2020:9201967. doi: 10.1155/2020/9201967. eCollection 2020. PMID 32099543
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884